CLINICAL TRIAL: NCT04374617
Title: Risk of Venous Thromboembolism in Critically Ill Patients With Severe COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)213/2020
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Critical Illness; Venous Thromboembolism; Venous Thromboses; Venous Thromboses, Deep; Venous Thrombosis Pulmonary; Pulmonary Embolism; Pulmonary Embolism and Thrombosis; Sars-CoV2; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Critical Illness; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Thrombosis; Severe Acute Respiratory Syndrome | interventions — Ultrasonography, Doppler, Duplex; Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Venous thromboembolism: Patients at risk of venous thromboembolism (deep venous thrombosis and/or pulmonary embolism)
  Interventions: Diagnostic Test: Duplex ultrasound and Computed Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Duplex ultrasound and Computed Tomography Angiography — All venous thromboembolisms suspected will diagnosed with ultrasound and CT-angiography
  Other Names: Compression ultrasound (CUS); Ct-Angiography

SUMMARY:
Severe COVID-19 patients at a high risk of venous thromboembolism. We studied patients in 2 intensive care units of university hospitals in Barcelona and Badalona, Spain. We performed a cut-off screening of deep venous thrombosis (DVT) with bilateral duplex ultrasound to 230 patients.

DETAILED DESCRIPTION:
SARS-CoV-2 infection has been associated with coagulation disorders and increased risk of venous thromboembolism (VTE). The aim of the study is to determine the cumulative incidence of VTE in critically ill patients with COVID-19 and its impact on prognosis.

Methods Cohort study of critically ill patients due to COVID-19. A bilateral venous compression (CUS) ultrasound screening of the lower extremities was performed during a cut-off period in 2 intensive care units of university hospitals in Spain. Asymptomatic and symptomatic VTE were registered: pulmonary embolism (PE) (diagnosed by CT-angiography) and deep venous thrombosis (DVT). The characteristics of the patients, results of their blood tests and their evolution after 7 days of follow-up were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe COVID-19 pneumonia admitted to the intensive care unit

Exclusion Criteria:

* Treatment with Extracorporeal membrane oxygenation (ECMO)
* Pregnant or postpartum women
* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe COVID-19 pneumonia admitted to the intensive care unit.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolisms | 7 days
  Patients with symptomatic pulmonary embolism confirmed on the CT-angiography and those with a swollen limb and confirmed deep venous thrombosis on compression ultrasound were considered to have "symptomatic venous thromboembolisms". The remaining patients with positive limb ultrasound or CT-angiography were considered to have "asymptomatic venous thrombembolism"

SECONDARY OUTCOMES:
Deaths | 7 days
  Deaths from all causes during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Bellmunt, MD,PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (3):
- Spain (3):
  - Vall d´Hebron Research Institute VHIR, Barcelona, Catalonia
  - Hospital Germans Trias i Pujol. Universitat Autònoma de Barcelona, Badalona
  - Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
We have planned to write a paper